CLINICAL TRIAL: NCT07215806
Title: A Phase I, Open-Label, Multiple-Dose Study of the Effect of Evobrutinib on the Pharmacokinetics of a Combined Oral Contraceptive in Healthy Female Participants
Brief Title: Effect of Evobrutinib on Pharmacokinetics of a Combined Oral Contraceptive
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MS200527_0079; 2022-000124-38 (EudraCT Number)
Record Dates: First submitted 2025-10-08; First posted 2025-10-14 (Actual); Results first posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Healthy
Keywords: Drug-drug interaction; Clinical pharmacology
MeSH Terms: interventions — Contraceptives, Oral, Combined; Ethinyl Estradiol; Norethindrone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COC + Evobrutinib (Experimental): Participants received combined oral contraceptive (COC) [0.03 milligrams (mg) of Ethinyl Estradiol (EE)], 0.5 mg of Norethisterone (NET)] orally on Day 1 and 15 in combination with Evobruitnib at a dose of 45 mg orally twice daily on Days 4 to 17.
  Interventions: Drug: Evobruitnib; Drug: Combined oral contraceptive [ethinyl estradiol/ norethisterone (EE/NET)]

INTERVENTIONS:
Drug: Evobruitnib — Participants received Evobruitnib at a dose of 45 mg orally twice daily on Days 4 to 17.
Drug: Combined oral contraceptive [ethinyl estradiol/ norethisterone (EE/NET)] — Participants received combined oral contraceptive (COC) [0.03 milligrams (mg) of Ethinyl Estradiol (EE)], 0.5 mg of Norethisterone (NET)] orally on Day 1 and 15.

SUMMARY:
The purpose of this study was to assess the effect of M2951 on the pharmacokinetics (PK) of a combined oral contraceptive [Ethinyl estradiol/Norethisterone (EE/NET)] in healthy female participants.

* Study Duration: up to 46 days
* Treatment Duration: Days 4 to 17 (14 days treatment with M2951); Days 1 and 15 (2 days treatment with Combined Oral Contraceptive [COC])
* Visit Frequency: Participants were resident in the Clinical Research Unit from Day -1 to Day 18.

ELIGIBILITY:
Inclusion Criteria:

* Participants are overtly healthy as determined by medical evaluation, including no clinically significant abnormality identified on physical examination or laboratory evaluation and no active clinically significant disorder, condition, infection or disease that would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion
* Participants have a body weight within 50.0 and 100.0 kilograms (kg) (inclusive) and body mass index within the range 19.0 and 30.0 kilograms per square meter (kg/m^2) (inclusive)
* Participants are nonsmokers for at least 6 months preceding Screening
* Female participants who are not a Woman of Childbearing Potential (WOCBP)
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participants with history or presence of clinically relevant respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders, as determined by medical evaluation
* Participants with diagnosis of hemochromatosis, Wilson´s disease, alpha 1 antitrypsin deficiency, or any other chronic liver disease including Gilbert's disease will be excluded from the study
* Participants with prior history of splenectomy or any clinically relevant surgery within 3 months prior to Screening
* Participants with history of any malignancy
* Participants with history of chronic or recurrent acute infection or any bacterial, viral, parasitic, or fungal infections within 30 days prior to Screening and at any time between Screening and admission, or hospitalization due to infection within 6 months prior to Screening
* Participants with history of shingles within 12 months prior to Screening
* Administration of live vaccines or live-attenuated virus vaccines within 3 months prior to Screening. Administration of other types of vaccines [e.g., Severe acute respiratory syndrome coronavirus 2 (SARSCoV2) vaccines] is allowed until 4 weeks before admission to CRU, thereafter it is prohibited until the end of the study
* Note: In case of clinical symptoms, the participant should be symptom-free for at least 1 week prior to admission to Clinical Research Unit (CRU)
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 68 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2022-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website http://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200527_0079
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | COC + Evobrutinib
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | COC + Evobrutinib
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Ethinyl Estradiol and Norethisterone
Description: AUC0-inf was calculated by combining AUC0-t and AUCextra. AUCextra represents an extrapolated value obtained by Clast pred/Lambda z, where Clast pred was the calculated serum concentration at the last sampling time point at which the measured serum concentration is at or above the Lower Limit of quantification (LLOQ) and Lambda z was the apparent terminal rate constant determined by log-linear regression analysis of the measured serum concentrations of the terminal log-linear phase.
Time Frame: Pre-dose, 0.3, 0.6, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60 and 72 hours post-dose on Days 1, 2, 3, 4, 15, 16, 17 and 18
Population: Pharmacokinetics (PK) Analysis set included all participants who have completed the study without any relevant protocol deviations and factors likely to affect the comparability of PK results; with adequate study intervention compliance; with evaluable PK data, i.e., no missing values for primary endpoints at each PK profile/assessment day (Day 1, Day 15).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour × picogram per milliliter (h×pg/mL)
Arm/Group | COC + Evobrutinib
Number analyzed (Participants) | 20
hour × picogram per milliliter (h×pg/mL)
  Ethinyl Estradiol | 1090 (26.7)
  Norethisterone | 36000 (35.9)

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Ethinyl Estradiol and Norethisterone
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | COC + Evobrutinib
Number analyzed (Participants) | 20
pg/mL
  Ethinyl Estradiol | 51.8 (30.1)
  Norethisterone | 4620 (34.0)

3. Secondary Outcome: Number of Participants With Treatment- Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether considered related to the study intervention or not. A serious AE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs were defined as events with onset date or worsening during the on-treatment period. TEAEs included both serious and non-serious TEAEs.
Time Frame: Up to 46 days
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | COC + Evobrutinib
Number analyzed (Participants) | 20
Participants | 9

4. Secondary Outcome: Number of Participants With Treatment- Emergent Adverse Events (TEAEs) by Severity
Description: The Investigator assessed the severity of each AE and SAE reported during the study and assign it to one of the following categories: Mild: An event that is easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities; Moderate: An event that causes sufficient discomfort and interferes with normal everyday activities; Severe: An event that prevents normal everyday activities. Do not confuse an AE that is assessed as severe with a SAE. Severe is a category used to rate the intensity of an event; both AEs and SAEs can be assessed as severe.
Time Frame: Up to 46 days
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | COC + Evobrutinib
Number analyzed (Participants) | 20
Participants
  Mild | 8
  Moderate | 1
  Severe | 0

5. Secondary Outcome: Change From Baseline in Hematology Parameter: Hemoglobin at Day 18
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the hematology parameter: hemoglobin.
Time Frame: Baseline, Day 18
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | COC + Evobrutinib
Number analyzed (Participants) | 20
gram per liter (g/L) | -8.780 (7.7256)

6. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes at Day 18
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the hematology parameter: Erythrocytes.
Time Frame: Baseline, Day 18
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | COC + Evobrutinib
Number analyzed (Participants) | 20
10^12 cells per liter | -0.29 (0.263)

7. Secondary Outcome: Change From Baseline in Hematology Parameters: Platelets, Leukocytes, Neutrophils, Eosinophils, Basophils, Monocytes and Lymphocytes at Day 18
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the hematology parameters: Platelets, Leukocytes, Neutrophils, Eosinophils, Basophils, Monocytes and Lymphocytes.
Time Frame: Baseline, Day 18
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | COC + Evobrutinib
Number analyzed (Participants) | 20
10^9 cells per liter
  Platelets | -18 (38.0)
  Leukocytes | -0.08 (1.395)
  Neutrophils | -0.21 (1.390)
  Eosinophils | -0.00 (0.050)
  Basophils | 0.00 (0.017)
  Monocytes | -0.02 (0.110)
  Lymphocytes | 0.16 (0.338)

8. Secondary Outcome: Change From Baseline in Hematology Parameters: Hematocrit, Basophils/Leukocytes, Eosinophils/Leukocytes, Lymphocytes/Leukocytes, Monocytes/Leukocytes and Neutrophils/Leukocytes at Day 18
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the hematology parameters: Hematocrit, Basophils/Leukocytes, Eosinophils/Leukocytes, Lymphocytes/Leukocytes, Monocytes/Leukocytes and Neutrophils/Leukocytes.
Time Frame: Baseline, Day 18
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | COC + Evobrutinib
Number analyzed (Participants) | 20
percentage of cells
  Hematocrit | -0.029 (0.0227)
  Basophils/Leukocytes | 0.0 (0.30)
  Eosinophils/Leukocytes | 0.0 (0.63)
  Lymphocytes/Leukocytes | 3.2 (8.44)
  Monocytes/Leukocytes | -0.2 (1.34)
  Neutrophils/Leukocytes | -3.0 (9.30)

9. Secondary Outcome: Change From Baseline in Coagulation Parameter: Activated Partial Thromboplastin Time at Day 18
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the coagulation parameter: Activated Partial Thromboplastin Time.
Time Frame: Baseline, Day 18
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | COC + Evobrutinib
Number analyzed (Participants) | 20
seconds | -1.6 (0.84)

10. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin at Day 18
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the hematology parameter: Erythrocytes Mean Corpuscular Hemoglobin.
Time Frame: Baseline, Day 18
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: picogram
Arm/Group | COC + Evobrutinib
Number analyzed (Participants) | 20
picogram | -0.06283 (0.541316)

11. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Volume at Day 18
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the hematology parameter: Erythrocytes Mean Corpuscular Volume.
Time Frame: Baseline, Day 18
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: femtoliters
Arm/Group | COC + Evobrutinib
Number analyzed (Participants) | 20
femtoliters | -0.7 (0.95)

12. Secondary Outcome: Change From Baseline in Coagulation Parameter: Prothrombin Intl. Normalized Ratio at Day 18
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the coagulation parameter: Prothrombin Intl. Normalized Ratio.
Time Frame: Baseline, Day 18
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | COC + Evobrutinib
Number analyzed (Participants) | 20
ratio | -0.02 (0.042)

13. Secondary Outcome: Change From Baseline in Chemistry Parameters: Bilirubin, Creatinine and Urate at Day 18
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the chemistry parameter: bilirubin, creatinine and urate.
Time Frame: Baseline, Day 18
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: micromole per liter (mcmol/L)
Arm/Group | COC + Evobrutinib
Number analyzed (Participants) | 20
micromole per liter (mcmol/L)
  Bilirubin | -0.8 (3.11)
  Creatinine | -4 (6.2)
  Urate | 4.1 (31.48)

14. Secondary Outcome: Change From Baseline in Chemistry Parameters: Aspartate Aminotransferase, Alanine Aminotransferase, Alkaline Phosphatase, Amylase, Lipase, Gamma Glutamyl Transferase and Lactate Dehydrogenase at Day 18
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the chemistry parameter: Aspartate Aminotransferase, Alanine Aminotransferase, Alkaline Phosphatase, Amylase, Lipase, Gamma Glutamyl Transferase and Lactate Dehydrogenase.
Time Frame: Baseline, Day 18
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | COC + Evobrutinib
Number analyzed (Participants) | 20
units per liter (U/L)
  Aspartate Aminotransferase | -2 (6.2)
  Alanine Aminotransferase | 3 (11.8)
  Alkaline Phosphatase | -4 (10.1)
  Amylase | -1 (7.5)
  Lipase | -2.0 (7.77)
  Gamma Glutamyl Transferase | 0 (5.4)
  Lactate Dehydrogenase | -35 (19.7)

15. Secondary Outcome: Change From Baseline in Chemistry Parameters: Sodium, Potassium, Calcium, Glucose, Chloride and Triglycerides at Day 18
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the chemistry parameter: Sodium, Potassium, Calcium, Glucose, Chloride and Triglycerides.
Time Frame: Baseline, Day 18
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | COC + Evobrutinib
Number analyzed (Participants) | 20
millimoles per liter (mmol/L)
  Sodium | 1 (2.6)
  Potassium | -0.03 (0.397)
  Calcium | -0.04 (0.077)
  Glucose | -0.10 (0.385)
  Chloride | 2 (2.4)
  Triglycerides | 0.2 (0.29)

16. Secondary Outcome: Change From Baseline in Chemistry Parameters: Total Protein at Day 18
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the chemistry parameter: Total Protein.
Time Frame: Baseline, Day 18
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | COC + Evobrutinib
Number analyzed (Participants) | 20
gram per liter (g/L) | -2 (3.5)

17. Secondary Outcome: Change From Baseline in Chemistry Parameters: C Reactive Protein at Day 18
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the chemistry parameter: C Reactive Protein.
Time Frame: Baseline, Day 18
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: milligram per liter (g/L)
Arm/Group | COC + Evobrutinib
Number analyzed (Participants) | 20
milligram per liter (g/L) | 4 (8.2)

18. Secondary Outcome: Change From Baseline in Vital Signs: Systolic Blood Pressure and Diastolic Blood Pressure at Day 18
Description: Diastolic blood pressure and systolic blood pressure were measured after at least 5 minutes of rest for the participant in a quiet sitting without distractions.
Time Frame: Baseline, Day 18
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | COC + Evobrutinib
Number analyzed (Participants) | 20
millimeters of mercury (mmHg)
  Systolic Blood Pressure | 4 (12.5)
  Diastolic Blood Pressure | 3 (9.7)

19. Secondary Outcome: Change From Baseline in Vital Signs: Pulse Rate at Day 18
Description: Pulse rate was measured after at least 5 minutes of rest for the participant in a quiet sitting without distractions.
Time Frame: Baseline, Day 18
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | COC + Evobrutinib
Number analyzed (Participants) | 20
beats per minute | 4 (10.6)

20. Secondary Outcome: Change From Baseline in Vital Signs: Respiratory Rate at Day 18
Description: Respiratory rate was measured after at least 5 minutes of rest for the participant in a quiet sitting without distractions.
Time Frame: Baseline, Day 18
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | COC + Evobrutinib
Number analyzed (Participants) | 20
breaths per minute | 0 (1.5)

21. Secondary Outcome: Change From Baseline in Vital Signs: Temperature at Day 18
Description: Temperature was measured after at least 5 minutes of rest for the participant in a quiet sitting without distractions.
Time Frame: Baseline, Day 18
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | COC + Evobrutinib
Number analyzed (Participants) | 20
degree Celsius | 0.2 (0.49)

22. Secondary Outcome: Change From Baseline in Electrocardiograms (ECGs) Parameter: Heart Rate at Day 18
Description: Heart rate was measured after at least 5 minutes of rest for the participant in a quiet sitting without distractions
Time Frame: Baseline, Day 18
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | COC + Evobrutinib
Number analyzed (Participants) | 20
beats per minute | -4 (7.5)

23. Secondary Outcome: Change From Baseline in Electrocardiograms (ECGs) Parameter: RR Duration, QT Duration, QTcF Duration, PR Duration, QRS Duration at Day 18
Description: RR Duration, QT Duration, QTcF Duration, PR Duration, QRS Duration was measured after at least 5 minutes of rest for the participant in a quiet sitting without distractions.
Time Frame: Baseline, Day 18
Population: Safety (SAF) analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | COC + Evobrutinib
Number analyzed (Participants) | 20
milliseconds (msec)
  RR Duration | 51 (98.4)
  QT Duration | 3 (17.8)
  QTcF Duration | -5 (11.0)
  PR Duration | 3 (15.3)
  QRS Duration | -2 (9.6)

24. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Ethinyl Estradiol and Norethisterone
Description: Time to reach the maximum observed plasma concentration (Tmax) was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 1
Population: Pharmacokinetics (PK) Analysis set included all participants: who have completed the study without any relevant protocol deviations and factors likely to affect the comparability of PK results; with adequate study intervention compliance; with evaluable PK data, i.e., no missing values for primary endpoints at each PK profile/assessment day (Day 1, Day 15).
Measure: Median (Full Range); unit: hours
Arm/Group | COC + Evobrutinib
Number analyzed (Participants) | 20
hours
  Ethinyl Estradiol | 3.00 [1.50 to 6.02]
  Norethisterone | 2.00 [0.667 to 3.00]

25. Secondary Outcome: Terminal Half Life (T1/2) of Ethinyl Estradiol and Norethisterone
Description: Terminal half-life was calculated as log2 divided by lambda z. Lambda z was terminal elimination rate constant determined from the terminal slope of the log-transformed plasma concentration curve.
Time Frame: as for outcome 1
Population: as for outcome 24
Measure: Median (Full Range); unit: hours
Arm/Group | COC + Evobrutinib
Number analyzed (Participants) | 20
hours
  Ethinyl Estradiol | 21.5 [10.5 to 32.1]
  Norethisterone | 12.7 [7.58 to 20.9]

26. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-t) of Ethinyl Estradiol and Norethisterone
Description: The AUC from time zero (= dosing time) to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification (LLOQ). Calculated using the mixed log-linear trapezoidal rule (linear up, log down).
Time Frame: as for outcome 1
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h×pg/mL
Arm/Group | COC + Evobrutinib
Number analyzed (Participants) | 20
h×pg/mL
  Ethinyl Estradiol | 964 (26.9)
  Norethisterone | 35100 (36.4)

27. Secondary Outcome: Apparent Total Body Clearance (CL/f) of Ethinyl Estradiol and Norethisterone
Description: Apparent total body clearance of drug from plasma following extravascular administration, calculated as dose/AUC0-infinity for Ethinyl Estradiol/Norethisterone.
Time Frame: as for outcome 1
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | COC + Evobrutinib
Number analyzed (Participants) | 20
Liter per hour
  Ethinyl Estradiol | 27.6 (26.7)
  Norethisterone | 13.9 (35.9)

28. Secondary Outcome: Apparent Volume of Distribution During Terminal Phase (VZ/f) of Ethinyl Estradiol and Norethisterone
Description: Vz/f is defined as the apparent volume of distribution during the terminal phase following extravascular administration for Ethinyl Estradiol/Norethisterone.
Time Frame: as for outcome 1
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | COC + Evobrutinib
Number analyzed (Participants) | 20
Liter
  Ethinyl Estradiol | 816 (26.0)
  Norethisterone | 252 (46.7)

ADVERSE EVENTS:
Time Frame: Up to 46 days
Arm/Group | COC + Evobrutinib
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 9/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COC + Evobrutinib (N=20)
Abnormal faeces (Gastrointestinal disorders) | 1 (1)
Defaecation urgency (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Restless legs syndrome (Nervous system disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 6 (6)
Polymenorrhoea (Reproductive system and breast disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT07215806/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-13): https://cdn.clinicaltrials.gov/large-docs/06/NCT07215806/SAP_001.pdf